CLINICAL TRIAL: NCT04382430
Title: Ultrasound Axillary Vein Access: Evaluation of Learning Curve for an Alternative Approach to Cardiac Device Implantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Seth Sheldon, Clinical Assistant Professor of Medicine - Cardiology, Principal Investigator, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00145717
Record Dates: First submitted 2020-05-03; First posted 2020-05-11 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Ultrasound Therapy; Complications; Cardiac Device Implant; Venous Access
Keywords: US Guided Venous access

STUDY DESIGN:
Intervention Model Description: The Study Group for this study will include 1 US experienced Electrophysiology (EP) attending, 4 US inexperienced EP attendings, and 1 US inexperienced EP fellow performing US cardiac device implantation (CDI). Each provider will perform 5 conventional CDI, 2 assisted US CDI to learn the procedure (except for experienced US attending), and 10 solo US CDI for a total of 17 procedures per provider (15 for experienced US attending). 100 patients will be needed for this study. This study will take approximately 16 weeks to complete.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- US Guided Axillary venous access (Experimental): Physician/ provider will perform 2 unassisted & 10 solo Ultrasound (US) guided venous access and pocket creation cardiac device implant. First 2 device implant will be done to educate physicians about ultrasound guided venous access. Subsequent subject will be randomized to 2:1 in ultrasound vs. conventional technique.
  Interventions: Procedure: Ultrasound guided venous access
- Conventional technique (Active Comparator): Physician/ provider will perform 5 cardiac device implant using conventional technique for venous access and pocket creation.
  Interventions: Procedure: Conventional technique

INTERVENTIONS:
Procedure: Ultrasound guided venous access — Each physician/ provider will perform 2 assisted ultrasound (US) guided venous access and pocket creation for cardiac device implant and 10 solo ultrasound guided cardiac device implant.
  Arms: US Guided Axillary venous access
Procedure: Conventional technique — Physician will perform 5 cardiac device implant using conventional technique of venous access and pocket creation
  Arms: Conventional technique

SUMMARY:
The purpose of this study is to determine the learning curve associated with Ultrasound (US) guided axillary vein access for cardiac device implantation based on length of procedure among operators of various levels of experience and to assess the 30-day complication rate for patients undergoing US guided device placement versus traditional implant methods.

DETAILED DESCRIPTION:
Ultrasound (US) guided axillary vein access for device implantation is an uncommon approach to gain venous access for cardiac device implantation - an extremely common procedure. However, there has been a growing trend of utilizing this approach to obtain venous access for device implantation among operators. Axillary vein access was described back as far as 1997, when it was utilized for contrast guided venipuncture to access the axillary vein for device implantation. Literature has suggested that an axillary venous approach, with either a superficial landmark or radiographic contrast, has better long-term efficacy and lower lead complications than a conventional subclavian approach for patients that had permanent pacemaker implantation. There are a variety of ways to access the axillary vein including contrast venography to help localization, "blind puncture" (utilizing fluoroscopy to identify anatomical landmarks), and US. More recently, operators have begun to utilize US guidance for axillary vein access. Esmaiel has described that US guidance for axillary vein access could potentially improve the success rate of venous access and limit complications. Others, albeit few, have reported US guided access for cardiac device implantation has the ability to reduce complications, is faster to complete, and easier to learn. According to the Agency for Healthcare Research and Quality in the United States, US guided central venous catheter placement is one of the 11 patient safety practices that have the strongest evidence supporting its use in improving patient outcomes. Evidence supports US guidance being standard of care in central venous catheter placement and using US for axillary access as helpful in cardiac device implantation, but providers still utilize predominantly alternative approaches to obtain venous access via the subclavian vein, cephalic cutdown, extrathoracic axillary using fluoroscopy and thoracic axillary using fluoroscopy.

Currently, there is limited data describing outcomes, the efficiency of US guided axillary access for cardiac device implantation, and the learning curve associated with this technique. Data suggests that utilizing the US approach can improve outcomes, be more efficient, and be easier to learn. Investigators recently reported a high success (95%) and low complication rate with US guided axillary access in 187 patients. Despite this limited data, operators still largely use alternative approaches for venous access. In part, this may be due to the learning curve associated with US axillary venous access.

While there is data demonstrating the utility of US guided axillary access, there is little evidence showing the learning curve for operators associated with this technique. The aim of this project is to assess the learning curve of this technique among operators of various levels of experience.

ELIGIBILITY:
Inclusion Criteria:

* Sign written Informed Consent Form.
* ≥18 years of age up to 90 years old.
* Eligible and referred for cardiac device implantation.
* BMI < 35.

Exclusion Criteria:

* Unable to sign consent.
* Patient eligible for cardiac device upgrades/ extractions, subcutaneous implantable cardioverter defibrillators (SICD) & leadless devices.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2021-06-06 (Actual); Study Completion 2021-06-06 (Actual)

PRIMARY OUTCOMES:
Venous access time between US guided and conventional technique | During procedure
  Assess changes in venous access and pocket creation time with progressive experience with US guided axillary venous access (learning curve).
Time spent for pocket creation between US guided venous access technique and conventional technique. | During procedure
  Compare the pocket creation time with US guided axillary venous access versus conventional techniques.
Time spent to obtain venous access & pocket creation between experienced and inexperienced physicians. | During procedure
  Compare venous access and pocket creation time amongst experienced and inexperienced physicians.
To assess 30 day post procedure complications | 30 Day post procedure
  Assess 30-day complications between techniques.
Assess acute procedural success between two techniques. | During procedure
  Compare overall procedural success whether device was successfully placed or not post procedure between US guided axillary venous access & conventional technique. Success as Assigned- whether implant technique assigned was successful or whether had to switch to an alternative technique.

CONTACTS AND LOCATIONS:
Overall Officials: Seth Sheldon, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramza BM, Rosenthal L, Hui R, Nsah E, Savader S, Lawrence JH, Tomaselli G, Berger R, Brinker J, Calkins H. Safety and effectiveness of placement of pacemaker and defibrillator leads in the axillary vein guided by contrast venography. Am J Cardiol. 1997 Oct 1;80(7):892-6. doi: 10.1016/s0002-9149(97)00542-0. PMID 9382004
- [Background] Kim KH, Park KM, Nam GB, Kim DK, Oh M, Choi H, Hong TJ, Park BM, Seo GW, Song PS, Kim DK, Seol SH, Kim DI, Kim YH, Choi KJ. Comparison of the axillary venous approach and subclavian venous approach for efficacy of permanent pacemaker implantation. 8-Year follow-up results. Circ J. 2014;78(4):865-71. doi: 10.1253/circj.cj-13-0884. Epub 2014 Mar 3. PMID 24583974
- [Background] Squara F, Tomi J, Scarlatti D, Theodore G, Moceri P, Ferrari E. Self-taught axillary vein access without venography for pacemaker implantation: prospective randomized comparison with the cephalic vein access. Europace. 2017 Dec 1;19(12):2001-2006. doi: 10.1093/europace/euw363. PMID 28064251
- [Background] Esmaiel A, Hassan J, Blenkhorn F, Mardigyan V. The Use of Ultrasound to Improve Axillary Vein Access and Minimize Complications during Pacemaker Implantation. Pacing Clin Electrophysiol. 2016 May;39(5):478-82. doi: 10.1111/pace.12833. Epub 2016 Mar 23. PMID 26880272
- [Background] Jones DG, Stiles MK, Stewart JT, Armstrong GP. Ultrasound-guided venous access for permanent pacemaker leads. Pacing Clin Electrophysiol. 2006 Aug;29(8):852-7. doi: 10.1111/j.1540-8159.2006.00451.x. PMID 16923001
- [Background] Seto AH, Jolly A, Salcedo J. Ultrasound-guided venous access for pacemakers and defibrillators. J Cardiovasc Electrophysiol. 2013 Mar;24(3):370-4. doi: 10.1111/jce.12005. Epub 2012 Nov 6. PMID 23131025
- [Background] Lin J, Adsit G, Barnett A, Tattersall M, Field ME, Wright J. Feasibility of ultrasound-guided vascular access during cardiac implantable device placement. J Interv Card Electrophysiol. 2017 Oct;50(1):105-109. doi: 10.1007/s10840-017-0273-3. Epub 2017 Jul 27. PMID 28752227
- [Background] Liccardo M, Nocerino P, Gaia S, Ciardiello C. Efficacy of ultrasound-guided axillary/subclavian venous approaches for pacemaker and defibrillator lead implantation: a randomized study. J Interv Card Electrophysiol. 2018 Mar;51(2):153-160. doi: 10.1007/s10840-018-0313-7. Epub 2018 Jan 15. PMID 29335840